CLINICAL TRIAL: NCT00646269
Title: Efficacy Assessment of Three Non Pharmacological Therapies in Alzheimer's Disease
Acronym: ETNA3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Caisse Nationale de Solidarité pour l'Autonomie (Other); National Health Insurance Fund for Unemployed Workers (Other); Direction Générale de la Santé, France (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Université Victor Segalen Bordeaux 2 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007/17
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Alzheimer's Disease
Keywords: Dementia ; Alzheimer's Disease ; Non pharmacological treatments ; cognitive training ; reminiscence therapy ; efficacy assessment
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator)
  Interventions: Behavioral: Standard intervention protocol
- 2 (Experimental)
  Interventions: Behavioral: Standard intervention protocol + Cognitive training therapy
- 3 (Experimental)
  Interventions: Behavioral: Standard intervention protocol + Reminiscence therapy
- 4 (Experimental)
  Interventions: Behavioral: Standard intervention protocol + "Made-to-measure" program

INTERVENTIONS:
Behavioral: Standard intervention protocol — The control group involves a standardized medical follow-up of patients with Alzheimer's disease and a psychoeducative group program for caregivers of patients.
  Arms: 1
Behavioral: Standard intervention protocol + Cognitive training therapy — "Cognitive training therapy" is provided in small groups of 5 to 8 patients. It consists in classroom type sessions designed to provide general cognitive stimulation. A set of standard cognitive exercises (involving memory, attention, or problem-solving…) related to activities of daily living is realized at each session.
  Arms: 2
Behavioral: Standard intervention protocol + Reminiscence therapy — "Reminiscence therapy" is provided in small groups of 5 to 8 patients. This therapy involves the discussion of past activities, events and experiences enhanced by aids such as photographs, familiar items, songs, or personal recordings. A particular topic of life (i.e. a wedding) is discussed at each session.
  Arms: 3
Behavioral: Standard intervention protocol + "Made-to-measure" program — The "made to measure" program involves no systematic intervention. The psychologist is asked to choose among the two possible therapies ("Cognitive training therapy" or "Reminiscence therapy") the one more suitable for the patient after considering his clinical characteristics including socio-demographic characteristics, disease severity or cognitive and behavioural disturbance. It is an individualized approach emphasizing the importance of flexibility to allow adjustment to individual needs.
  Arms: 4

SUMMARY:
ETNA3 is a multicentric randomised clinical trial conducted in France to evaluate the impact of cognitive training, reminiscence therapy and a "made-to-measure" program on the progression rate of dementia.

DETAILED DESCRIPTION:
ETNA3 is a multicentric randomised clinical trial conducted in France to evaluate the impact of non pharmacological treatments on the progression rate of dementia: Three non pharmacological treatments are being studied: cognitive training therapy, reminiscence therapy and a "made-to-measure" program. Nearly 40 "Memory Clinics" are participating. 800 patients suffering Alzheimer's Disease in the mild to moderate stage of the disease will be included. For each therapy, a standard intervention protocol has been defined. The main objective is to determine whether any or several of these non pharmacological treatments can delay the severe stage of dementia during a 2-year follow-up. The secondary outcomes assess cognitive abilities, functional abilities in activities of daily living, behavioural disturbance, apathy, quality of life, depression, caregiver burden and resource utilization

ELIGIBILITY:
Inclusion Criteria:

* Patients in the mild to moderate stages of Alzheimer's Disease : MMSE score between 16 and 26 ; and stages 3 to 5 of the Global Deterioration Scale
* Patients over 50 years of age
* Patients with social security affiliation

Exclusion Criteria:

* Patients suffering other type of dementia
* Institutionalized patients
* Patients with psychiatric disorder
* Patients with severe pathology in the terminal stages
* Patients receiving non pharmacological therapies other than that proposed in the study
* Enrollment in a pharmacological trial in the first 6 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Proportion of progression to the severe stage of Alzheimer's disease (MMSE score of 15 or lower) | 2 years

SECONDARY OUTCOMES:
Cognitive abilities (ADAS-cog) | 2 years
Functional abilities in activities of daily living (DAD scale) | 2 years
Behavioural disturbance (NPI) | 2 years
Apathy (Apathy Inventory) | 2 years
Quality of life (Quol-AD) | 2 years
Depression (MADRS) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François, Dartigues, MD, PhD, Principal Investigator — University Hospital, Bordeaux; Geneviève Chêne, MD, PhD, Study Chair — University Hospital, Bordeaux
Locations (39):
- France (39):
  - CH Agen, Agen
  - CHU Amiens Nord, Amiens
  - Centre Mémoire de Ressources et de Recherches de Bordeaux, CHU de Bordeaux, Bordeaux
  - Hôpital Pellegrin, Bordeaux
  - CHU Côte de Nacre, Caen
  - Centre pour Personnes Agées, Colmar
  - Centre de Gériatrie, Dax
  - Hôpital Dupuytren, Draveil
  - Pôle de Gérontologie CHICAS, Gap
  - Les Fontaines de Monjous, Gradignan
  - CMRR & Neuropsychologie, Pavillon de Neurologie, CHU de Grenoble, Grenoble
  - Centre Hospitalier La Rochelle, La Rochelle
  - Association AA83 Alzheimer Aidants Var Etablissement " Les pensées ", La Seyne-sur-Mer
  - Centre Hospitalier de Libourne, Libourne
  - CHU Limoges, Limoges
  - Hôpital Privé Gériatrique Les Magnolias, Longjumeau
  - Centre Hospitalier Bretagne Sud, Lorient
  - Groupe Hospitalier Saint-Augustin, Malestroit
  - Hôpital Sainte-Marguerite, Marseille
  - Centre Antonin Balmes, Montpellier
  - Hôpital Gui de Chauliac, Montpellier
  - Clinique Neurologique, CHU Nord, Nantes
  - Centre Mémoire, Hôpital Pasteur,, Nice
  - Hôpital Broca, Paris
  - Hôpital de la Salpétrière,, Paris
  - Centre Hospitalier des Pyrénées, Pau
  - Hôpital de Jour Gériatrique, Pau
  - Hôpital Xavier-Arnozan, Pessac
  - CHI Poissy-saint-germain-en-laye, Poissy
  - Hôpital de Jour gériatrique, Poitiers
  - CHU de Rennes, Rennes
  - CHRU de Saint-Etienne, Saint-Etienne
  - Centre hospitalier Ariège Couserans, Saint-Girons
  - Hôpital de Jour Gériatrique, Saint-Raphaël
  - Hôpitaux universitaires de Strasbourg, Strasbourg
  - Bagatelle, Talence
  - CHIC Marmande - Tonneins, Tonneins
  - CHU Purpan-Casselardit, Toulouse
  - Hôpital des Charpennes, Villeurbanne

REFERENCES:
- [Background] Clare L, Woods RT, Moniz Cook ED, Orrell M, Spector A. Cognitive rehabilitation and cognitive training for early-stage Alzheimer's disease and vascular dementia. Cochrane Database Syst Rev. 2003;(4):CD003260. doi: 10.1002/14651858.CD003260. PMID 14583963